CLINICAL TRIAL: NCT00107575
Title: Improving Smoking Cessation Outcomes in Heavy Drinkers
Brief Title: Improving Smoking Cessation Outcomes in Heavy Drinkers - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Christopher W. Kahler, Professor, Brown University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: NIDA-15534-1; R01-15534-1
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Results first posted 2010-01-11 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-09

CONDITIONS: Tobacco Use Disorder
Keywords: tobacco; alcohol
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Ethanol; Methods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard treatment (ST) (Active Comparator): Standard smoking cessation treatment (ST)
  Interventions: Other: Standard treatment (ST)
- ST-BI (Experimental): Standard treatment plus a brief alcohol intervention
  Interventions: Behavioral: Standard treatment plus brief alcohol intervention

INTERVENTIONS:
Behavioral: Standard treatment plus brief alcohol intervention — Standard smoking cessation treatment with nicotine patch plus a brief alcohol-focused intervention
  Arms: ST-BI
Other: Standard treatment (ST) — Behavioral smoking cessation counseling and nicotine patch.
  Arms: Standard treatment (ST)

SUMMARY:
To test the effectiveness of an smoking cessation treatment for smokers who also drink alcohol heavily.

DETAILED DESCRIPTION:
Heavy alcohol use frequently co-occurs with cigarette smoking and may impede smoking cessation. This clinical trial examined whether smoking cessation treatment that incorporates brief alcohol intervention can improve smoking cessation outcomes (7-day verified point prevalence abstinence) and reduce drinks consumed per week. Heavy drinkers seeking smoking cessation treatment were assigned by urn randomization to receive, along with 8-weeks of nicotine replacement therapy, either a 4-session standard smoking cessation treatment (ST, n = 119) or standard treatment of equal intensity that incorporated brief alcohol intervention (ST-BI, n = 117).

ELIGIBILITY:
Inclusion Criteria:

1. be at least 18 years of age
2. have smoked cigarettes regularly for at least one year
3. currently smoke at least 10 cigarettes a day
4. currently be using no other tobacco products or nicotine replacement therapy
5. currently drink heavily according to self-report (>14 drinks per week or >5 drinks per occasion at least once per month over the last 12 months for men; >7 drinks per week or >4 drinks per occasion at least once per month over the past 12 months for women)

Exclusion Criteria:

1. meet full DSM-IV criteria for alcohol dependence in the past 12 months
2. meet criteria for other current psychoactive substance abuse or dependence (excluding nicotine dependence and alcohol abuse) in the past 12 months [this would also exclude individuals with lifetime substance dependence who continue to have some abuse/dependence symptoms in the past 12 months]
3. meet criteria for current dysthymia, major depression, or manic episode [past month]
4. are currently psychotic [past 12 months] or suicidal [suicidal ideation or intent in the past month]
5. have an unstable medical condition that would suggest caution in the use of the nicotine patch (e.g., unstable angina pectoris, arrhythmia, recent congestive heart failure)
6. are currently pregnant or lactating or intend to become pregnant. We also will exclude participants who are not alcohol dependent but who have characteristics that might make supervised alcohol detoxification necessary (e.g., morning drinking to avoid withdrawal, daily drinking of >12 drinks, recent withdrawal symptoms, history of severe withdrawal symptoms such as hallucinations, seizures, or delirium tremens).

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2003-08; Primary Completion 2007-06 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W Kahler, Ph.D., Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

REFERENCES:
- [Result] Kahler CW, Metrik J, LaChance HR, Ramsey SE, Abrams DB, Monti PM, Brown RA. Addressing heavy drinking in smoking cessation treatment: a randomized clinical trial. J Consult Clin Psychol. 2008 Oct;76(5):852-62. doi: 10.1037/a0012717. PMID 18837602

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Treatment: Standard smoking cessation treatment (ST) including 4 sessions of behavioral counseling and nicotine patch
- Standard Treatment Plus a Brief Alcohol Intervention (ST-BI): Standard treatment of 4 individual behavior counseling sessions and nicotine patch, with treatment also incorporating brief alcohol intervention
Period: Overall Study
Arm/Group | Standard Treatment | Standard Treatment Plus a Brief Alcohol Intervention (ST-BI)
Started | 119 | 117
Completed | 108 | 107
Not Completed | 11 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Treatment | Standard Treatment Plus a Brief Alcohol Intervention (ST-BI) | Total
Number analyzed (Participants) | 119 | 117 | 236
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 2
  Between 18 and 65 years | 113 | 112 | 225
  >=65 years | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (12.1) | 42.3 (11.8) | 41.5 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 53 | 106
  Male | 66 | 64 | 130
Region of Enrollment [Number; unit: participants]
  United States | 119 | 117 | 236

OUTCOME MEASURES:

1. Primary Outcome: Smoking Abstinence at 26 Weeks
Description: 7 days of smoking abstinence confirmed biochemically at 26 week post quit attempt
Time Frame: 26 weeks
Population: For analyses of smoking outcomes, missing data were considered smoking. However, at 26 weeks, 2 participants in ST-BI had died and therefore their data was left as missing for this period.
Measure: Number; unit: participants
Arm/Group | Standard Treatment | Standard Treatment Plus a Brief Alcohol Intervention (ST-BI)
Number analyzed (Participants) | 119 | 115
participants | 21 | 22
Statistical Analysis 1: Comparison: Standard Treatment vs Standard Treatment Plus a Brief Alcohol Intervention (ST-BI); Test type: Superiority or Other; p > .05, Chi-squared

2. Secondary Outcome: Alcohol Drinks Consumed Per Week Over a 2-week Period
Description: Average number of standard alcoholic drinks consumed per week over each 2-week period across the 26 weeks of follow-up as assessed by the Timeline Followback Interview. Standard alcoholic drink is defined as 12 oz of beer, 5 oz of wine, or 1.5 ounces of liquor.
Time Frame: At 2, 8, 16, and 26-week follow-ups
Population: The number of participants analyzed reflects the number of participants who provided at least some valid data on the Timeline Followback Interview
Measure: Mean (Standard Deviation); unit: drinks
Arm/Group | Standard Treatment | Standard Treatment Plus a Brief Alcohol Intervention (ST-BI)
Number analyzed (Participants) | 106 | 110
drinks
  Drinks per week: Weeks 1-2 | 9.8 (10.0) | 8.2 (9.9)
  Drinks per week: Weeks 3-4 | 10.3 (10.4) | 8.4 (10.8)
  Drinks per week: Weeks 5-6 | 10.3 (10.9) | 9.1 (11.1)
  Drinks per week: Weeks 7-8 | 10.7 (10.7) | 9.6 (11.2)
  Drinks per week: Weeks 9-10 | 10.1 (9.7) | 9.1 (9.8)
  Drinks per week: Weeks 11-12 | 9.5 (9.8) | 9.2 (10.3)
  Drinks per week: Weeks 13-14 | 10.5 (11.2) | 8.6 (9.1)
  Drinks per week: Weeks 15-16 | 10.6 (11.0) | 9.2 (9.6)
  Drinks per week: Weeks 17-18 | 10.9 (10.3) | 9.0 (10.3)
  Drinks per week: Weeks 19-20 | 10.8 (10.3) | 9.8 (11.8)
  Drinks per week: Weeks 21-22 | 10.1 (9.3) | 9.1 (11.2)
  Drinks per week: Weeks 23-24 | 9.8 (8.6) | 9.1 (12.0)
  Drinks per week: Weeks 25-26 | 10.9 (9.9) | 10.0 (13.3)
Statistical Analysis 1: Comparison: Standard Treatment vs Standard Treatment Plus a Brief Alcohol Intervention (ST-BI); Test type: Superiority or Other; p = .027, generalized estimating equations — a priori p-value was p < .05; Negative binomial model controlling for sex, motivation to change drinking, and baseline drinking; expected count ratio = 0.81, 95% CI 2-sided [0.67 to 0.98]

3. Primary Outcome: Smoking Abstinence at 16 Weeks
Description: 7 days of smoking abstinence confirmed biochemically at 16 weeks
Time Frame: 16 weeks
Measure: Number; unit: Participants
Arm/Group | Standard Treatment | Standard Treatment Plus a Brief Alcohol Intervention (ST-BI)
Number analyzed (Participants) | 119 | 117
Participants | 21 | 21
Statistical Analysis 1: Comparison: Standard Treatment vs Standard Treatment Plus a Brief Alcohol Intervention (ST-BI); Test type: Superiority or Other; p = .18, Chi-squared

4. Primary Outcome: Smoking Abstinence at 8 Weeks
Description: 7 days of smoking abstinence confirmed biochemically at 8 weeks
Time Frame: 8 weeks
Measure: Number; unit: Participants
Arm/Group | Standard Treatment | Standard Treatment Plus a Brief Alcohol Intervention (ST-BI)
Number analyzed (Participants) | 119 | 117
Participants | 37 | 46
Statistical Analysis 1: Comparison: Standard Treatment vs Standard Treatment Plus a Brief Alcohol Intervention (ST-BI); Test type: Superiority or Other; p = .95, Chi-squared

5. Primary Outcome: Smoking Abstinence at 2 Weeks
Description: 7 days of smoking abstinence confirmed biochemically at 2 weeks
Time Frame: 2 weeks
Measure: Number; unit: Participants
Arm/Group | Standard Treatment | Standard Treatment Plus a Brief Alcohol Intervention (ST-BI)
Number analyzed (Participants) | 119 | 117
Participants | 54 | 67
Statistical Analysis 1: Comparison: Standard Treatment vs Standard Treatment Plus a Brief Alcohol Intervention (ST-BI); Test type: Superiority or Other; p = .76, Chi-squared

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Standard Treatment | Standard Treatment Plus a Brief Alcohol Intervention (ST-BI)
Serious Adverse Events (participants affected / at risk) | 0/119 | 2/117
Other Adverse Events (participants affected / at risk) | 0/119 | 0/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Treatment (N=119) | Standard Treatment Plus a Brief Alcohol Intervention (ST-BI) (N=117)
Death (General disorders) | 0 | 2
Lung Cancer (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No